CLINICAL TRIAL: NCT03424811
Title: Mobile Health (mHealth) Nutrition Intervention for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 827786
Record Dates: First submitted 2018-01-10; First posted 2018-02-07 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Diet Modification

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Includes core behavior change strategies and behavioral skills training designed to promote healthy eating behaviors.
  Interventions: Device: Mobile Health Intervention
- Control Group (No Intervention): Information provided will mimic what families may receive during a routine well-child visit.

INTERVENTIONS:
Device: Mobile Health Intervention — Mobile health intervention to promote healthy eating.
  Arms: Intervention Group

SUMMARY:
The high prevalence of mealtime difficulties and obesity among children with autism spectrum disorder (ASD) calls for new and innovative ways to promote healthy eating and weight development in this population. This project aims to develop and test an interactive mobile health (mHealth) nutrition intervention, which incorporates core behavior change strategies that have been empirically tested in family-based nutrition research and behavioral interventions with children with ASD. The feasibility and efficacy of this mHealth intervention to improve dietary outcomes in children with ASD will be tested in a proof-of-concept randomized controlled trial.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is the fastest growing developmental disability affecting more than 2 million US children and tens of millions worldwide. Children with ASD are 5 times more likely to have mealtime challenges and be picky eaters, which in part has been attributed to restrictive and ritualistic behaviors and heightened sensory sensitivity. These nutritional difficulties pose significant every day challenges for caregivers when it comes to child feeding and daily eating routines and call for new and innovative ways to promote healthy eating in children affected by ASD. The use of mobile technologies is rapidly increasing in children across all age groups. Children with ASD, in particular, often engage with mobile devices on a daily basis and mobile health (mHealth) technology has been shown to be an effective tool for improving behavioral, social, and communication skills in children with ASD. The investigators aim to harness the lure of technology and develop and test, for the first time, the feasibility and acceptability of an interactive mHealth nutrition intervention for children with ASD. This intervention will build upon core behavior change strategies that have been empirically tested in family-based nutrition research for over 3 decades. A second aim of this project is to test, in a 3-month randomized controlled trial, the efficacy of the mHealth intervention on changing consumption of targeted healthy and less healthy foods and beverages in 6- to 10-year-old children with ASD who are picky eaters. Primary outcomes of this proof-of-concept trial will include 3-month changes in children's daily intake of fruits and vegetables, salty and sugary snacks, and sugar-sweetened beverages. Secondary outcomes will include parent and child engagement with the mHealth technology, motivation, user friendliness and ease of use. If successful, the use of this innovative mHealth nutrition intervention will offer new and powerful targets for intervention in improving dietary intake and the fight against childhood obesity in this especially vulnerable population of children.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 10 years;
* fluent in English;
* have an ASD diagnosis;
* cognitive skills within average (or higher) range with IQ ≥ 80;
* above or standardized receptive language scores.

Exclusion Criteria:

* moderate-severe hearing/visual or motor impairment;
* taking antipsychotic medications;
* on special diet;
* are underweight (BMI-for-age < 5th percentile).

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kuschner, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Slater CN, Schroeder K, Fultz A, Kuschner ES, O'Malley L, Johnson K, Benvenuti T, Chittams J, Quinn RJ, Graham Thomas J, Pinto-Martin J, Levy SE, Kral TVE. Insights from user experience and evaluation of a mobile health nutrition intervention for children with autism: A qualitative study. J Hum Nutr Diet. 2024 Dec;37(6):1439-1453. doi: 10.1111/jhn.13365. Epub 2024 Sep 9. PMID 39248190
- [Derived] Kral TVE, O'Malley L, Johnson K, Benvenuti T, Chittams J, Quinn RJ, Thomas JG, Pinto-Martin JA, Levy SE, Kuschner ES. Effects of a mobile health nutrition intervention on dietary intake in children who have autism spectrum disorder. Front Pediatr. 2023 Feb 15;11:1100436. doi: 10.3389/fped.2023.1100436. eCollection 2023. PMID 36873654

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started (Baseline) | 19 | 19
Completed (3-month Follow-Up) | 10 | 19
Not Completed | 9 | 0
Not completed — Lost to Follow-up | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.9 (1.2) | 8.4 (1.4) | 8.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 12 | 17 | 29
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 11 | 15 | 26
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 1
Child BMI-for-age-percentile [Mean (Standard Deviation); unit: percentile] | 68.1 (34.2) | 63.1 (37.2) | 65.6 (35.4)

OUTCOME MEASURES:

1. Primary Outcome: 3-month Fruit and Vegetable Intake
Description: 24-hour dietary recalls to assess fruit and vegetable intake
Time Frame: Change from baseline intake of fruits and vegetables at 3 months
Measure: Mean (Standard Error); unit: Servings per day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 19
Servings per day | 2.16 (0.43) | 3.01 (0.41)

2. Primary Outcome: 3-month Snack Intake
Description: 24-hour dietary recalls
Time Frame: Change from baseline intake to end of intervention (3 months)
Measure: Mean (Standard Error); unit: Calories per day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 19
Calories per day | 420.8 (58.4) | 385.7 (51.0)

3. Primary Outcome: 3-month Sugar-sweetened Beverage Intake
Description: 24-hour dietary recalls to assess sugar-sweetened beverage intake.
Time Frame: Change from baseline to end of intervention (3 months)
Measure: Mean (Standard Error); unit: Fluid ounces per day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 19
Fluid ounces per day | 7.6 (1.7) | 7.3 (1.6)

4. Secondary Outcome: Evaluation of mHealth Intervention - User Evaluation
Description: The study aimed to better understand participant experiences with motivation, user-friendliness, ease of use of the mobile health technology.
Time Frame: 3 months
Population: Feedback from caregivers in the intervention group.
Measure: Number; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 10
Participants
  Number of parents who said app was helpful for increasing child's consumption of healthy foods. | 4
  Number of parents who said app was helpful for decreasing child's consumption of unhealthy foods. | 2

5. Secondary Outcome: Evaluation of mHealth Intervention - Technology Engagement
Description: Parents in the intervention group will be asked to complete a semi-structured interview, which will ask them about parent and child engagement with the technology.
Time Frame: 3 months
Population: Feedback from caregivers in the intervention group.
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 10
participants
  Number of parents who said that they enjoyed using the app somewhat or very much. | 7
  Number of parents who said that their child enjoyed using the app somewhat or very much. | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the entire 3-month intervention period.
Description: Adverse event collection followed the definition from clinicaltrials.gov
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
The coronavirus pandemic significantly interfered with the conduct of the study. All home visits had to be stopped in March of 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03424811/Prot_SAP_000.pdf